CLINICAL TRIAL: NCT00636220
Title: Evaluation of the DPP HIV Test With Reader and the HIV 1/2 Stat-Pak Test Using Oral Fluids
Brief Title: Evaluation of the DPP HIV 1/2 Test and the HIV 1/2 Stat Pak Test Using Oral Fluid
Acronym: HIVOF
Status: Completed | Type: Observational
Sponsor: Chembio Diagnostic Systems, Inc. (Industry)
Collaborators: University of Maryland (Other)
Responsible Party: Sponsor
Other Study IDs: P-HIV-01; UMB Protocol # H-29110
Record Dates: First submitted 2008-03-10; First posted 2008-03-14 (Estimated); Results first posted 2010-02-15 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-07

CONDITIONS: HIV Infections
Keywords: HIV-1 Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — oral fluid samples and venous blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- A, Observational

SUMMARY:
This protocol is intended to test the feasibility of using the HIV 1/2 STAT-PAK and the DPP HIV 1/2 test (with and without the DPP Handheld Reader) to detect HIV antibodies in oral fluids.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the feasibility of using fresh oral fluid specimens, from known HIV-positive individuals, to test for HIV-1 antibodies using both the DPP HIV 1/2 and HIV 1/2 STAT-PAK tests. Two oral fluid collection devices will be used and compared (MPC and Chembio collection devices) and the results obtained from oral fluids will be compared with those obtained from whole blood and plasma using paired samples from the same participants. The comparison between oral fluid, whole blood and plasma will be made in both Chembio devices (HIV 1/2 STAT-PAK and DPP HIV 1/2).

ELIGIBILITY:
Inclusion Criteria:

* Participants with known HIV infection who are willing to participate in the study and who sign an informed consent (or assent), will be included in the study.
* Patients on HAART treatment for HIV will be included, but this information as well as the dates (duration) of treatment will be obtained through the interview of study participants; a medical record review is not necessary or required. The study participant's responses will be recorded by study staff on a Data Collection Form.
* Patients with immunosuppressive conditions other than HIV will be included if available, but will be limited to < 25% of the total test population. Immunosuppression will also be assessed through interview of study participants and/or through verbal confirmation by the treating physician; a medical record/chart review is not required.
* Patients must be willing to undergo venipuncture to donate one tube of EDTA whole blood (not more than 10cc), and to provide three oral fluid samples.

Exclusion Criteria:

* Patients who do not consent, withdraw consent, or for whom the investigator determines that venipuncture or gum swabbing may create a health risk will be excluded from the study.
* Participants who have been enrolled in HIV vaccine studies will be excluded from the study. This will be ascertained through interview of study participants.
* Participants who have been enrolled once in this study will be excluded from repeat enrollment.
* Participants must not have introduced any substance into their oral cavity (gum, food, beverage, candy, lozenges, mouthwash, etc.) for 30 minutes prior to providing an oral fluid sample. This will be ascertained through interview of study participants.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of 100 participants with known (clinically or serologically) confirmed HIV infection. The participants, recruited by the staff of the Laboratory of Vial Diagnostics from the Evelyn Jordan Center, may be males or females (including pregnant women) at least 12 years of age from any ethnic and racial background.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2008-03; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Niel Constantine, PhD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- Evelyn Jordan Center, University of Maryland, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment time period was from March 13, 2008 to July 1, 2008. All enrollment was at the Evelyn Jordan Center, University of Maryland Baltimore (UMD).
Groups:
- Confirmed HIV Infection: The study population will consist of 100 participants with known (clinically or serologically) confirmed HIV infection.
Period: Overall Study
Arm/Group | Confirmed HIV Infection
Started | 101
Completed | 101
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Confirmed HIV Infection: participants with known (clinically or serologically) confirmed HIV infection.
Arm/Group | Confirmed HIV Infection
Number analyzed (Participants) | 101
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 101
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 60
Region of Enrollment [Number; unit: participants]
  United States | 101
Fresh Oral Fluid Samples with known HIV reactivity [Number; unit: samples] — Fresh Oral Fluid samples were collected from participants with known HIV+ status. HIV reactivity was clinically or serologically confirmed.
  samples | 101
Participants with known HIV reactivity [Number; unit: Participants] — participants with known HIV reactivity
  Participants | 101

OUTCOME MEASURES:

1. Primary Outcome: Number of Fresh Oral Fluid Samples With Known HIV (+) Status and HIV Reactivity
Description: Known HIV status determined clinically or serologically. HIV reactivity for all 100 samples determined first by licensed EIA and then confirmed with Western Blot and/or NAT testing.
Time Frame: 1 to 3 days
Measure: Number; unit: samples
Arm/Group | Confirmed HIV Infection
Number analyzed (Participants) | 100
samples | 100

2. Secondary Outcome: The Effectiveness of MPC and Chembio Oral Fluid Collection Devices
Time Frame: 1-3
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Confirmed HIV Infection
Serious Adverse Events (participants affected / at risk) | 0/100
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No